CLINICAL TRIAL: NCT05673304
Title: Immune and Pathological Response in Breast Cancer After Preoperative Irradiation With Stereotactic Technique and Neoadjuvant ChemOtherapy
Brief Title: Preoperative Boost Associated With Neoadjuvant Chemotherapy in Luminal B Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBISCO Trial
Record Dates: First submitted 2023-01-04; First posted 2023-01-06 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer; Radiotherapy
Keywords: Luminal B Breast Cancer; Neoadjuvant radiation therapy; Neoadjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): Patients will be treated on the primary tumour with a total dose of 24 Gy (8 Gy x 3 fractions QD) within 2 weeks from the start of neoadjuvant chemotherapy
  Interventions: Radiation: SBRT anticipated boost
- observational cohort (No Intervention): This cohort will include patients fulfilling inclusion criteria who refuse enrollment in the interventional cohort and patients where SBRT boost appears not feasible after enrollment for technical issues

INTERVENTIONS:
Radiation: SBRT anticipated boost — 24 Gy in 3 fractions to the tumour
  Arms: Interventional group

SUMMARY:
IBISCO TRIAL is a phase II trial aimed to demonstrate the improvement of pathological complete response (pCR) in Luminal B breast cancer (BC) patients treated with stereotactic radiation therapy (SBRT) as an anticipated boost associated with neoadjuvant chemotherapy (NAC).

As a secondary objective, histochemical and molecular analysis of the tumour and the inflammatory microenvironment will be performed.

DETAILED DESCRIPTION:
IBISCO TRIAL is a phase II trial aimed to demonstrate the improvement of pCR in Luminal B breast cancer (BC) patients treated with stereotactic radiation therapy (SBRT) as an anticipated boost associated with neoadjuvant chemotherapy (NAC).

The primary endpoint will be evaluated on surgical specimen using the residual cancer burden (RCB) index.

Thirty patients with clinical stage T1-2 Luminal B BC, suitable for conservative surgery and with a clinical indication for NAC, will be enrolled in two years. An observation cohort will also be created with patients fulfilling inclusion criteria who refuse enrollment in the interventional cohort and for patients where SBRT boost appears not feasible after enrollment for technical issues.

As a secondary objective, histochemical and molecular analysis of the tumour and the inflammatory microenvironment will be performed.

After the completion of neoadjuvant treatments, surgery and adjuvant therapies (endocrine therapy and whole breast irradiation) will be performed as for clinical practice

ELIGIBILITY:
Inclusion Criteria:

* Luminal B-like BC, cT1-2
* Indication for neoadjuvant chemotherapy

Exclusion Criteria:

* Pregnancy
* Breast feeding
* Patient not available for follow up

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
pCR | 6 month after SBRT (at surgery)
  pathological complete response rate (according to AJCC-TNM and RCB) after SBRT anticipated boost

SECONDARY OUTCOMES:
acute toxicity | immediate to 6 months after SBRT
  acute toxicity after SBRT, evaluated according to CTCAE v.5
late toxicity | from 6 months after SBRT
  late toxicity after completion of treatments (included adjuvant RT), evaluated according to CTCAE v.5

CONTACTS AND LOCATIONS:
Overall Officials: Alessio G Morganti, MD, PhD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No